CLINICAL TRIAL: NCT03996174
Title: What Are the Palliative Care Needs of the Mahoran Population Take Into Consideration the Socio-anthropological Specificities of This Population, But Also the Demographic, Social, Health and Geographical Characteristics of Mayotte Island
Brief Title: Palliative Care Needs Assessment of the Population Living in Mayotte (French Island of Comoros)
Acronym: SP-MAYOTTE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2019/430
Record Dates: First submitted 2019-06-03; First posted 2019-06-24 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-05

CONDITIONS: Palliative Therapy
Keywords: Palliative care; needs assessment; Mayotte; terminal care
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Interview — Interview bases on the use of an interview guide, during one hour maximum

SUMMARY:
This qualitative study aims to explore the assessment of palliative care needs of the population living in Mayotte, French territory of the Comoros.

The aim is to offer a palliative care service tailored to the needs of the population in this area.

ELIGIBILITY:
Inclusion Criteria:

* patients study: to be at the palliative stage of his illness, informed consent
* family study: being a family or caregiver of a patient in palliative care, informed consent
* care workers study: being a care worker of a patient in palliative care, informed consent

Exclusion Criteria:

* 0

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 3 studies will be conducted: one with "palliative patients" identified by their care workers, one with their family or caregivers, and one with their care workers.
  .
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
individual semi-structured interviews | day 1
  individual semi-structured interviews to obtain a aata saturation
  Reliability and Validity of the research described according to Guba.

CONTACTS AND LOCATIONS:
Overall Officials: Régis Aubry, MD, PhD, Study Director — Service douleur, soins palliatifs
Locations (1):
- CHRU Besançon, Besançon, France